CLINICAL TRIAL: NCT01459432
Title: A Study to Evaluate the Persistence of Antibody Seven Years After a Booster Dose of Either a Glycoconjugate or a Polysaccharide Vaccine Against Serogroup C Neisseria Meningitidis Given to Adolescents
Brief Title: Understanding Immunity Persistence After Adolescent MenC Vaccination
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OVG 2011/03
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Antibody Persistance After Booster Dose of Men C Vaccine
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Follow-on blood sample from previous study
  Interventions: Other: Venepuncture and blood sample collection.

INTERVENTIONS:
Other: Venepuncture and blood sample collection. — Venepuncture and blood sample collection.

SUMMARY:
The main purpose of this study is to evaluate the duration of immunity after a booster dose of a MenC-CRM vaccine given to adolescents between 13 and 15 years of age. Does seroprotection persist beyond teenage years and into the early twenties? This is the age group which is most likely to carry the organism and to transmit it to other members of the population. If a booster dose of MenC vaccine given to adolescents does produce protective levels of antibody which persist into early adulthood, this would strengthen the case for such a booster to be added to the UK routine immunisation schedule, to reduce the risk of a resurgence of the disease in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed clinical study M14P2E1
* Participant who are willing to participate and who would be expected to comply with the requirements of the protocol
* Participants who have given informed consent for participation in the study

Exclusion Criteria:

* History of invasive meningococcal C disease (or any case of invasive meningococcal disease where the serotype was unknown)
* Confirmed or suspected immunosuppressive or immunodeficient conditions, including human immunodeficiency virus (HIV) infection
* Severe blood clotting disorders

Ages: 20 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults, approximately 20 - 23 years old.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with rSBA titre ≥1:8 (correlate of protection). | 4 months

SECONDARY OUTCOMES:
Geometric mean titre (GMT) rSBA. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Vaccine Group, Oxford, United Kingdom

REFERENCES:
- [Derived] de Whalley PC, Snape MD, Plested E, Thompson B, Nuthall E, Omar O, Borrow R, Pollard AJ. Long-term seroprotection after an adolescent booster meningococcal serogroup C vaccination. Arch Dis Child. 2013 Sep;98(9):686-91. doi: 10.1136/archdischild-2013-303893. Epub 2013 Jul 13. PMID 23853000